CLINICAL TRIAL: NCT05634967
Title: Post-Authorization Safety Study for Assessment of Pregnancy and Infant Outcomes in Patients Treated With Kesimpta (Ofatumumab) Using OTIS Observational Pregnancy Surveillance Program and DMSKW Registry
Brief Title: Kesimpta (Ofatumumab) Pregnancy Registry
Status: Recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: COMB157G2403
Record Dates: First submitted 2022-11-22; First posted 2022-12-02 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Multiple Sclerosis; Pregnancy
Keywords: PASS; Kesimpta; ofatumumab; Pregnancy; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — ofatumumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Disease-matched cohort (Comparison Group 1): comparison group consisting of women diagnosed with MS who have not used Kesimpta during pregnancy (unexposed disease-matched comparison group).
- Healthy cohort (only applicable in the Kesimpta-OTIS sub-study) (Comparison Group 2): healthy women who are not diagnosed with MS or any other autoimmune disease, have not had exposure to a known human teratogen, and have not taken Kesimpta in pregnancy (healthy comparison group). Since the DMSKW register is an MS population specific register that does not collect data on non-MS population, this cohort is only applicable in the Kesimpta-OTIS sub-study.
- Kesimpta-exposed cohort: women and infants who are exposed to Kesimpta during pregnancy to treat MS.
  Interventions: Other: Kesimpta

INTERVENTIONS:
Other: Kesimpta — Prospective non-interventional study. There is no treatment allocation. Patients participating in from the two independent sub-studies, namely the Kesimpta-OTIS sub-study and Kesimpta-DMSKW sub-study, of identical design, conducted in parallel, enrolling pregnant women (MS and non-MS) residing in US or Canada and pregnant women (MS only) from Germany respectively are eligible for enrolling to this study.
  Other Names: Ofatumumab
  Groups: Kesimpta-exposed cohort

SUMMARY:
The Kesimpta Pregnancy Registry is an observational, exposure cohort designed study to examine pregnancy and infant outcomes in women and infants who are exposed to Kesimpta (ofatumumab) during pregnancy to treat MS.

DETAILED DESCRIPTION:
The study is expected to enroll for approximately 7 years and follow the pregnant women and their infant(s) over a maximum of 21 months.

The study will be conducted as two sub-studies leveraging independent ongoing pregnancy registries:

* The Organization of Teratology Information Specialists (OTIS) Research Group, University of California, San Diego, USA (referred to as "OTIS") will serve as data source for the Kesimpta-OTIS sub-study;
* The German MS and pregnancy registry - Deutschsprachigen Multiple Sklerose und Kinderwunsch Register (DMSKW) at Katholisches Klinikum Bochum gGmbH, St Josef Hospital, Bochum, Germany (referred to as "DMSKW") will serve as data source for the Kesimpta- DMSKW sub-study.

Both registries will independently collect and assess data related to the pregnancy and infant outcomes of interest and provide aggregate data which will be further combined (metaanalyses) by Novartis (referred to as the Sponsor) or a designated contract research organization (CRO).

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all the criteria listed under the respective cohorts to enroll in that particular cohort of the registry:

Cohort 1: Kesimpta-Exposed Cohort

1. Pregnant women
2. Diagnosed with MS, with the indication validated by medical records when possible
3. Administered Kesimpta for the treatment of MS at any time from 166 days prior to the first day of the LMP, or up to and including the end of pregnancy
4. Agree to the conditions and requirements of the study including the interview schedule, release of medical records, the dysmorphology examination of live born infants (OTIS specific), and validated developmental performance questionnaire in live born children

Cohort 2: Disease-Matched Comparison Cohort (Comparison Group 1)

1. Pregnant women
2. Diagnosed with MS, with the indication validated by medical records when possible
3. May or may not have taken another medication for MS in the current pregnancy
4. Agree to the conditions and requirements of the study including the interview schedule, release of medical records, the dysmorphology examination of live born infants (OTIS specific), and validated developmental performance questionnaire in live born children

Cohort 3: Healthy Comparison Cohort (Comparison Group 2):Kesimpta-OTIS sub-study specific

1. Pregnant women
2. Agree to the conditions and requirements of the study including the interview schedule, release of medical records, the dysmorphology examination of live born infants, and validated developmental performance questionnaire in live born children

Exclusion Criteria:

Women meeting any of the following criteria will be excluded from the cohort study:

Cohort 1: Kesimpta-Exposed Cohort

1. Women who have enrolled in the Kesimpta cohort study with a previous pregnancy
2. Women who have used Kesimpta for an indication other than a currently approved indication
3. Women with exposure to any of the following medications within 5 half-lives (or pharmacodynamic effect when relevant) prior to conception:

   * Other anti-CD20 monoclonal antibody: same class as Kesimpta
   * S1P modulators: same class as Mayzent
   * Cladribine (Mavenclad): Based on the US label, animal studies indicate that there is positive evidence of teratogenicity for Cladribine
   * Teriflunomide (Aubagio): The teratogenecity of teriflunomide is unknown and currently under investigation.
   * New medications (marketed after 2021) indicated for the treatment of MS will be evaluated for inclusion/exclusion criteria as the study progresses.
4. Retrospective enrollment after the outcome of pregnancy is known (i.e. the pregnancy has ended prior to enrollment)
5. Results of diagnostic test(s) that are positive for a major structural defect prior to enrollment. However, women who have had any normal or abnormal prenatal screening or diagnostic test prior to enrollment are eligible as long as the test result does not indicate a major structural defect.

Cohort 2: Disease-Matched Comparison Cohort (Comparison Group 1)

1. Administered Kesimpta 166 days before the first day of LMP or anytime during pregnancy
2. Women with exposure to any of the following medications within 5 half-lives (or pharmacodynamic effect when relevant) of conception:

   * Anti CD-20 monoclonal antibody
   * Cladribine (Mavenclad)
   * S1P modulators
   * Teriflunomide (Aubagio) New medications (marketed after 2021) indicated for the treatment of MS will be evaluated for inclusion/exclusion criteria as the study progresses.
3. Women who have enrolled in the Kesimpta cohort or BAF312A2403 Mayzent cohort with a previous pregnancy
4. Retrospective enrollment after the outcome of pregnancy is known (i.e. the pregnancy has ended prior to enrollment)
5. Results of diagnostic test(s) that are positive for a major structural defect prior to enrollment. However, women who have had any normal or abnormal prenatal screening or diagnostic test prior to enrollment are eligible as long as the test result does not indicate a major structural defect.

Cohort 3: Healthy Comparison Cohort (Comparison Group 2): Only applicable to Kesimpta-OTIS sub-study

1. Administered Kesimpta 166 days before or Mayzent 4 days after the first day of LMP or anytime during pregnancy
2. Women who have a diagnosis of a MS
3. Women who have a current diagnosis of any autoimmune disease
4. Women who have first contact with the project after prenatal diagnosis of any major structural defect
5. Women treated with Mayzent or Kesimpta for non-MS indication
6. Retrospective enrollment after the outcome of pregnancy is known (i.e. the pregnancy has ended prior to enrollment)
7. Results of diagnostic test(s) that are positive for a major structural defect prior to enrollment. However, women who have had any normal or abnormal prenatal screening or diagnostic test prior to enrollment are eligible as long as the test result does not indicate a major structural defect.
8. Women exposed to a known human teratogenic drugs during pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women and their infant(s)
Study Population: Participants from sub-studies, namely the Kesimpta-OTIS sub-study and Kesimpta-DMSKW sub-study, of identical design, conducted in parallel, enrolling pregnant women (MS and non-MS) residing in US or Canada and pregnant women (MS only) from Germany respectively.
Sampling Method: Non-Probability Sample
Enrollment: 725 (Estimated)
Dates: Start 2023-01-05 (Actual); Primary Completion 2033-02-28 (Estimated); Study Completion 2033-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of participants with major structural defects | Up to 21 months
  Number of participants with major structural defects will be collected

SECONDARY OUTCOMES:
Number of participants with spontaneous abortion/miscarriage | Up to 21 months
  Number of participants with spontaneous abortion/miscarriage will be collected
Number of stillbirth cases | Up to 21 months
  Number of stillbirth cases will be collected
Number of elective termination cases | Up to 21 months
  Number of elective termination cases will be collected
Number of preterm delivery cases | Up to 21 months
  Number of preterm delivery cases will be collected
Number of preeclampsia / eclampsia cases | Up to 21 months
  Number of preeclampsia / eclampsia cases will be collected
Number of cases with pattern of 3 or more minor structural defects | Up to 21 months
  Number of cases with pattern of 3 or more minor structural defects will be collected
Number of participants small for gestational age | Up to 21 months
  Number of participants small for gestational age will be collected
Number of participants with postnatal growth small for age at one year of age | Up to 21 months
  Number of participants with postnatal growth small for age at one year of age will be collected
Developmental performance at approximately one year of age: Michaelis developmental milestones questionnaires | Up to 21 months
  The Michaelis developmental milestones questionnaires will be used to assess the developmental performance in live born infants.
Developmental performance at approximately one year of age: Denver developmental screening test | Up to 21 months
  Denver developmental screening test will be used to assess the developmental performance in live born infants;
Number of serious or opportunistic infections in the first year of life. | Up to 21 months
  Number of serious or opportunistic infections in the first year of life will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- University of California San Diego OTIS, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: MotherToBaby Pregnancy Studies are observational studies coordinated at the University of California San Diego. Our studies are currently enrolling pregnant women in a study examining the use of medications to treat multiple sclerosis during pregnancy. — https://mothertobaby.org/ongoing-study/kesimpta-ofatumumab/